CLINICAL TRIAL: NCT01932164
Title: Use of Mesenchymal Stem Cells for Alveolar Bone Tissue Engineering for Cleft Lip and Palate Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sirio-Libanes (Other)
Collaborators: Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other)
Responsible Party: Principal Investigator, Daniela Franco Bueno, DDS; PhD, Hospital Sirio-Libanes
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSL 2013-04
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Results first posted 2015-03-30 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Cleft Lip and Palate
Keywords: Cleft lip and palate; Deciduous dental pulp stem cells; mesenchymal stem cells; tissue engineering; bone tissue engineering; bioengineering
MeSH Terms: conditions — Cleft Lip | interventions — Alveolar Bone Grafting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cleft lip and palate (Experimental): 5 Patients with cleft unilateral lip and palate that have already performed the alignment of dental arches through the recommended orthodontic treatment will be selected to be submited to alveolar bone tissue engineering surgery
  Interventions: Procedure: maxillary alveolar graft by tissue engineering; Procedure: Bone tissue engineering using mesenchymal stem cells

INTERVENTIONS:
Procedure: maxillary alveolar graft by tissue engineering — Extraction of deciduous teeth of cleft lip and palate patients to obtain mesenchymal stem cells;
  Other Names: alveolar bone graft; bone tissue engineering; bone tissue engineering using mesenchymal stem cells
Procedure: Bone tissue engineering using mesenchymal stem cells — Secondary alveolar graft in patients with cleft lip and palate using using mesenchymal stem cell obtained from dental pulp of deciduous teeth (autogenous) associated with a biomaterial composed of collagen and hydroxyapatite.

SUMMARY:
The aim of this study is to perform the bone tissue engineering to reconstruct the alveolar bone defect in cleft lip and palate patients using mesenchymal stem cells from deciduous dental pulp associated with a collagen and hydroxyapatite biomaterial (Geistlich Bio-Oss®) through prospective qualitative and quantitative analysis of bone neoformation.

DETAILED DESCRIPTION:
The reconstruction of the craniofacial skeleton in development between 2 and 10 years old, remains a major challenge for reconstructive plastic surgery. Local autogenous bone is practically unavailable, the distant bone graft has significant morbidity and use of alloplastic materials is incompatible with the growing facial skeleton. With the advent of bioengineered tissue, however, osteogenesis induced by the use of mesenchymal stem cells associated with biomaterials has become a potential solution to the shortage bone-related morbidity and donor bone in the region in pediatric patients.

The association of mesenchymal stem cells to biomaterials has provided new bone formation and a significant reduction of morbidity, for rehabilitation of the alveolar bone in patients with cleft lip palate.

To perform the rehabilitation of alveolar bone cleft, other donor regions of bone (iliac crest, ribs, skull) suffer morbidity for obtaining bone to be used in alveolar bone grafting. In order to eliminate the morbidity at the bone donor region for these patients and reduce costs of patient permanence in the operating room the aim of this study is to perform the bone tissue engineering to reconstruct the alveolar bone defect in cleft lip and palate patients using mesenchymal stem cells from deciduous dental pulp associated with a collagen and hydroxyapatite biomaterial (Geistlich Bio-Oss®) through prospective qualitative and quantitative analysis of bone neoformation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unilateral cleft lip and palate ;
* Patient who has performed the treatment to align the dental arches in the ambulatory of odontology at Hospital Municipal Infantil Menino Jesus;
* Patient that have Goslow index 1, 2 or 3;
* Patiente which have 2/3 of the root of the canine tooth (cleft region) formed.

Exclusion Criteria:

* Prior alveolar surgery;
* Canine teeth erupted before the bone graft;
* Presence of co-morbidities;
* Incomplete documentation;
* Patients who have not done all the multidisciplinary treatment at Hospital Municipal Infantil Menino Jesus.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2015-12-16 (Actual); Study Completion 2015-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela F Bueno, PhD, Principal Investigator — Hospital Sírio-Libanês
Locations (1):
- Hospital Sírio Libanês, São Paulo, Brazil

REFERENCES:
- [Background] Hibi H, Yamada Y, Ueda M, Endo Y. Alveolar cleft osteoplasty using tissue-engineered osteogenic material. Int J Oral Maxillofac Surg. 2006 Jun;35(6):551-5. doi: 10.1016/j.ijom.2005.12.007. Epub 2006 Apr 11. PMID 16584868
- [Background] Gimbel M, Ashley RK, Sisodia M, Gabbay JS, Wasson KL, Heller J, Wilson L, Kawamoto HK, Bradley JP. Repair of alveolar cleft defects: reduced morbidity with bone marrow stem cells in a resorbable matrix. J Craniofac Surg. 2007 Jul;18(4):895-901. doi: 10.1097/scs.0b013e3180a771af. PMID 17667684
- [Derived] Tanikawa DYS, Pinheiro CCG, Almeida MCA, Oliveira CRGCM, Coudry RA, Rocha DL, Bueno DF. Deciduous Dental Pulp Stem Cells for Maxillary Alveolar Reconstruction in Cleft Lip and Palate Patients. Stem Cells Int. 2020 Mar 12;2020:6234167. doi: 10.1155/2020/6234167. eCollection 2020. PMID 32256610

RESULTS

PARTICIPANT FLOW:
Recruitment Details: the recruitment of 5 patients was performed at dentistry department of Hospital Menino Jesus between june and august 2013.
Groups:
- Cleft Lip and Palate: Patients with cleft unilateral lip and palate that have already performed the alignment of dental arches through the recommended orthodontic treatment
  maxillary alveolar graft by tissue engineering: Extraction of deciduous tooth of cleft lip and palate patients to obtain mesenchymal stem cells; Secondary graft by bone tissue engineering using mesenchymal stem cell obtained from dental pulp of deciduous teeth (autogenous) associated with a biomaterial composed of collagen and hydroxyapatite.
Period: Overall Study
Arm/Group | Cleft Lip and Palate
Started | 5 (It was performed the selection of 5 patients to participate of these study (08/2013))
Cleft Lip and Palate | 5 (It was performed de extraction of deciduous teeth of 5 cleft lip/palate patients (09/2013))
Cleft Lip and Palate | 5 (Dental pulp was obtained from teeth of 5 different patients (09/2013))
Cleft Lip and Palate | 5 (Mesenchymal stem cell obtained from dental pulp of 5patients was obtained, caractherized and frozen)
Cleft Lip and Palate | 5 (Alveolar bone graft surgeries were did using their dental pulp stem cells with biomaterial)
Cleft Lip and Palate | 5 (The surgeries were performed between december 2013 and june 2014.)
Completed | 5 (In all 5 patients we observed bone formation closing the alveolar cleft after 6 months)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cleft Lip and Palate
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — 3 female and 2 male children with cleft lip and palate were submited to bone tissue engineering alveolar bone graft.
  Participants
    Female | 3
    Male | 2
Region of Enrollment [Number; unit: participants]
  Brazil | 5

OUTCOME MEASURES:

1. Primary Outcome: Amount of New Bone Mass Formed
Description: The quantification of bone formation will be conducted by analysis of CT scans of alveolar cleft area that receive autogenous mesenchymal stem cells from dental pulp associated with the biomaterial 3 and 6 months after surgical procedure ( tissue engineering ) in comparison with CT Scan previously of tissue engineering surgery.Preoperative and follow-up examinations reveled progressive alveolar bone union in all patients. For these 5 patients final completion of the alveolar defect with an 89,5% mean bone height was detected 6 months postoperatively. We are still waiting the canine dental eruption at the new bone. For these group of patients the bone tissue engineering using autologous mesenchymal stem cells associated with biomaterial resulted in satisfactory bone healing.
Time Frame: 6 months from surgical procedure for alveolar grafting;
Population: 3 females and 2 males with cleft lip and palate
Measure: Mean (95% Confidence Interval); unit: percentage of bone formation
Arm/Group | Cleft Lip and Palate
Number analyzed (Participants) | 5
percentage of bone formation | 89 [89 to 100]

2. Primary Outcome: Quality of Bone Regeneration
Description: The quality of bone formation will be conducted by analysis of CT scans of alveolar cleft area through canine tooth eruption in these position of new bone formation by tissue engineering techniques. We are waiting the canine eruption at the mouth.
Time Frame: Three months after the graft
Measure: Mean (80% Confidence Interval); unit: percentage of bone filling
Arm/Group | Cleft Lip and Palate
Number analyzed (Participants) | 5
percentage of bone filling | 90 [80 to 100]

ADVERSE EVENTS:
Time Frame: The adverse event data were collected on days 15th, 1 month, 6 months and 12 months of all 5 patients.
Description: All adverse event information used by clinical trial were used.
Groups:
- Cleft Lip and Palate: 5 Patients with cleft unilateral lip and palate that have already performed the alignment of dental arches through the recommended orthodontic treatment
  maxillary alveolar graft by tissue engineering: Extraction of deciduous tooth of cleft lip and palate patients to obtain mesenchymal stem cells; Secondary graft by bone tissue engineering using mesenchymal stem cell obtained from dental pulp of deciduous teeth (autogenous) associated with a biomaterial composed of collagen and hydroxyapatite.
Arm/Group | Cleft Lip and Palate
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes